CLINICAL TRIAL: NCT03854357
Title: The Effect of Focused Rehabilitation on Subscapularis Strength After Total Shoulder Arthroplasty
Brief Title: Subscapularis Strength After Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Lafi Khalil, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12088
Record Dates: First submitted 2019-02-12; First posted 2019-02-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Osteoarthritis
Keywords: Subscapularis; Total Shoulder Arthroplasty; Subscapularis Rehabilitation; Subscapularis strength

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional Isolated Subscapularis Rehabilitation (Experimental): Patients will be randomized to receive additional isolated subscapularis specific rehabilitation exercises during their standard post-operative physical therapy sessions after anatomic total shoulder arthroplasty.
  Interventions: Procedure: Subscapularis Rehabilitation; Procedure: Standard Rehabilitation
- Standard Post-Operative TSA Rehabilitation (Active Comparator): Patients will be randomized to receive additional isolated subscapularis specific rehabilitation exercises during their standard post-operative physical therapy sessions after anatomic total shoulder arthroplasty.
  Interventions: Procedure: Standard Rehabilitation

INTERVENTIONS:
Procedure: Subscapularis Rehabilitation — Specific subscapularis rehabilitation exercises which are not included in the current, standard rehabilitation protocol assigned to total shoulder arthroplasty patients post-operatively.
  Arms: Additional Isolated Subscapularis Rehabilitation
Procedure: Standard Rehabilitation — Standard post-operative rehabiliation protocol assigned to all total shoulder arthroplasty patients postoperatively

SUMMARY:
This is a randomized, double-blinded, standard of care-controlled clinical trial. The purpose of this study is to determine the difference in subscapularis strength and function after anatomic Total Shoulder Arthroplasty (aTSA) in patients who receive isolated subscapularis rehabilitation in addition to the standard rehabilitation after surgery at 12-month follow up. Specifically the investigators will measure subscapularis strength utilizing a dynamometer device and subscapularis function utilizing isolated subscapularis physical examination testing: belly-press, bear-hug, and lift-off tests. Additionally, investigators will document secondary outcome measures including shoulder range of motion and Patient Reported Outcome Measure Information System (PROMIS) questionnaire scores.

DETAILED DESCRIPTION:
Study Design: This is a randomized, double-blinded, standard of care-controlled clinical trial. All adult patients undergoing anatomic total shoulder arthroplasty for glenohumeral osteoarthritis will be included and randomized after surgery into either the control group which is prescribed a standard rehabilitation protocol or the intervention group which also is prescribed the same standard rehabilitation protocol with the the addition of isolated subscapularis rehabilitation.

Purpose: To determine the subscapularis strength and function after anatomic total shoulder arthroplasty (aTSA) in patients who receive isolated subscapularis rehabilitation in addition to the standard rehabilitation protocol as compared to those who only receive the standard rehabilitation protocol at 12-month follow up. Specifically the investigators will measure subscapularis strength utilizing a dynamometer and subscapularis function utilizing isolated subscapularis physical examination testing: belly-press, bear-hug, and lift-off tests.

Hypothesis: The investigators believe that subscapularis strength can be improved using isolated subscapularis rehabilitation in addition to standard rehabilitation, leading to improved outcomes in patients receiving aTSA. This should also improve the post-operative physical examination predicting a functional subscapularis tendon.

Rationale and expectations: Anatomic total shoulder arthroplasty is often performed in patients with severe glenohumeral osteoarthritis that have an intact subscapularis. Often times it is seen that these patients return with positive isolated subscapularis tests, despite the subscapularis being intact after surgery. If these patients require revision surgery, an ultrasound is the only test that can be performed to evaluate the status of the subscapularis tendon. This study is difficult and not 100% accurate. It needs to be determined if the patient will need a reverse total shoulder arthroplasty due to the positive subscapularis test findings. Previous studies by Baumgartner et al. showed that patients that received a total shoulder arthroplasty with tenotomy improved liftoff, and bear-hug strength testing, but operative shoulder strength remained inferior to strength of the nonoperative shoulder. Patients with improvements in strength were more likely to have greater improvements in outcome scores and range of motion. It was noted that improvements in the shoulder activity level after anatomic total shoulder arthroplasty may be dependent on improvements in strength. The investigators believe that subscapularis strength can be improved using isolated subscapularis rehabilitation in addition to standard rehabilitation, leading to improved outcomes in patients receiving aTSA. This should also improve the post operative physical examination predicting a functional subscapularis tendon.

Research Plan: Patients to be included in the study will be those with glenohumeral osteoarthritis with an intact rotator cuff that are undergoing anatomic total shoulder arthroplasty. Exclusion criteris includes patients undergoing revision shouder arthroplasty, a previous subscpaularis rotator cuff repair or deficient rotator cuff, patients with inflammatory arthropathies, such as rheumatoid arthritis, and patients with a history of infection in the shoulder joint. Reverse total shoulder arthroplasty will be excluded. Non-English speaking patients will be excluded from the study in order to simplify communication with study participants. The control population will consist of patients undergoing the standard rehabilitation protocol for aTSA. Patients will be undergoing rehabilitation regardless of study participation.

Protocol and Technique:

Recruitment: Patients meeting inclusion criteria undergoing aTSA will be recruited and consented for participation in the study at their pre-operative clinic visit. Their pre-operative strength and function testing will occur at this time.

Randomization: Placement into the study group or control group will be randomized and prospectively followed. The randomization process will remain blinded to surgeon, patient, and all co-investigators except for the primary physical therapist lead in the project (lead PT). At the first post-operative visit within the first month post-operatively, the patient will receive a physical therapy prescription per standard protocol. At the time of physical therapy initiation, the lead PT in the project will contact the patient's physical therapist and provide them with instructions regarding the research study, including which group the patient has been randomized into (standard vs additional subscapularis rehab) and strict instructions to perform the physical therapy without informing the patient of their randomized assignment. Upon making contact with the physical therapist, the lead PT provides them with a manual with the exact rehabilitation protocol assigned to the patient, ensuring that regardless of which physical therapy the patient elects to undergo treatment by, they receive the same standard physical therapy, plus the same standard subscapularis rehabilitation exercises (if randomized into the study group).

Follow up testing: The post-operative strength and function of patients in both treatment groups, isolated subscapularis rehabilitation with standard rehabilitation and standard rehabilitation alone, will be measured at subsequent 3 months, 6 months and 12 month postoperative visits. Measurements taken are outlined above and include shoulder range of motion (forward flexion, abduction, abduction-erternal rotation, abduction-internal rotation, external rotation), ability to perform a belly press, lift off, and bear hug test. Strength for internal rotation and subscapularis strength will be performed, using the dynamometer.

Data: Patients will be asked to fill out questionnaires for this study at each time point (preoperative, postoperative at months 3, 6, and 12). These include PROMIS Bank v2.0 - Upper Extremity, PROMIS Bank v1.1 - Pain Interference, and ASES. Strength scores will be assessed using a Lafayette Manual Muscle Testing System Model 01165 (dynamometer) to measure peak force in lbs. The means of each group along with standard deviation will be calculated for each parameter measured. P-value of 0.05 will be utilized for statistically significant results.

Primary Endpoint: Strength (measured by dynamometer testing) of the subscapularis.

Secondary Endpoint: Function and outcomes as measured by range of motion and questionnaire scores of pain and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over the age of 18
* Must have a diagnosis of glenohumeral osteoarthritis
* Must be scheduled for primary anatomic total shoulder arthroplasty.

Exclusion Criteria:

* History of prior rotator cuff surgery
* Rotator cuff deficiency
* Planned reverse total shoulder arthroplasty
* inflammatory arthropathy
* prior shoulder replacement surgery
* neurologic deficits of the affected extremity
* diagnosis of frozen shoulder
* previous infection in the shoulder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Subscapularis Strength | 12 months post-operative follow-up
  Subscapularis strength is the single, primary outcome measure. It will be measured by a dynamometer device, which is a device that patient holds in their hand and presses against a static object (such as a wall), creating force which is measured by the device. The device records this force as pounds (lb). Therefore, the investigators will use the dynamometer device to measure the single, primary outcome measure of strength (of the subscapularis muscle), with the single output unit of "pounds of force" in order to measure changes in strength from pre-operative testing to post-operative testing (at 3, 6, and 12 month post-operative time points).

SECONDARY OUTCOMES:
Shoulder Range of Motion | 12 months post-operative follow-up
  Shoulder range of motion will be measured using a goniometer at all time points, to compare improvement in range of motion from preoperative to post-operative testing time points. A goniometer is a device which allows an investigator to measure a subject's range of motion of a limb or extremity using the unit of measure "degrees" in all planes of motion. Investigators will measure the range of motion of the subject's shoulder (upper extremity) in the following planes: forward flexion, abduction, external rotation, abduction external rotation, and abduction internal rotation. These will be compared from pre-operative baseline measurements through 12-month post-operative measurements.
Patient Reported Outcome Measure Information System | 12 months post-operative follow-up
  Patient reported outcomes will be collected through a series of questionnaires administered at each time point: preoperative, and 3, 6, and 12 month postoperative clinic visits. The investigators will administer the questionnaire to the subjects, which includes the Patient Reported Outcome Measurement Information System (PROMIS) outcome score questionnaire. The PROMIS scores from this questionnaire are scaled from a minimum score of 0 to a maximum score of 100, where 50 is the mean, and 10 is the standard deviation. The scores of the patients will be compared from baseline preoperative recordings through the 12-month post-operative follow up.
Subscapularis Function | 12 months post-operative follow up.
  Subscapularis function will be determined as either "intact" or "deficient" based on the clinical examination of the subscapularis muscle using functional provocative tests such as the belly press, bear hug, and lift off lag test for subscapularis function at each respective time point. These tests are clinical tests which investigators use in clinic to evaluate the ability of the subscapularis muscle to function. Depending on body habitus and shoulder range of motion, patients may be unable to perform some or all of these tests. For this reason, one test will be administered to any given patient, depending on which test they are able to perform. The outcome of the test will be reported as either an intact or a deficient subscapularis tendon function. Therefore this will account for one outcome measure of subscapularis function.

CONTACTS AND LOCATIONS:
Overall Officials: Lafi S Khalil, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided